CLINICAL TRIAL: NCT02569502
Title: Open Label, Nonrandomized Clinical Trial of Safety and Tolerability of Enfuviritide (Fuzeon®, HIV Fusion Inhibitor) in Patients With Advanced HIV1 Infection
Brief Title: A Study of Enfuvirtide (Fuzeon) in Patients With Advanced Human Immunodeficiency Virus-1 (HIV-1) Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18634
Record Dates: First submitted 2015-10-05; First posted 2015-10-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

ARMS (1):
- Enfuvirtide (Experimental): Participants will receive 180 milligrams (mg) of enfuvirtide adminstered twice daily as subcutaneous injections
  Interventions: Drug: enfuvirtide

INTERVENTIONS:
Drug: enfuvirtide — Participants will receive a total daily dose of 180mg of enfurtide administered twice daily as a subcutaneous injection.
  Other Names: Fuzeon

SUMMARY:
This study will evaluate the safety and tolerability of subcutaneous Fuzeon in patients with advanced HIV-1 infection unable to construct an appropriate treatment regimen from currently available antiretroviral agents. The anticipated time on study treatment is 3-12 months, and the target sample size is 9 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult or adolescent patients greater than (>)16 years of age
* HIV-1 infection
* CD4 count less than (<)350/cubic millimeters (mm^3)
* HIV RNA viral load >10,000 copies per milliliter (copies/mL) while on highly active antiretroviral therapy (HAART)
* Documented resistance, treatment-limiting toxicity, and/or >=6 months' prior experience with each of 3 currently available classes of antiretroviral drugs.

Exclusion Criteria:

* Women who are pregnant or breastfeeding;
* Patients unable to self-inject;
* Active, untreated opportunistic infection.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who discontinue enfuvirtide due to adverse events\n | Up to 102 weeks
Percentage ofparticipants who discontinue from tratment since they no longer wish to continue with the injections | Up to 102 weeks
Percentage of participants with Serious Adverse Events (SAEs) and Serious AIDS-Defining events | Up to 102 weeks

SECONDARY OUTCOMES:
Percentage os participants reporting serious adverse events on the first day of study dosing and up to 28 days after discontinuiation of the study drug | Up to 28 days after discontinuation of enfuvirtide
Percentage of participants with Injection Site Reactions (ISR) and who discontinued enfuvirtide due to ISR | Up to 102 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (1):
- Sofia, Bulgaria